CLINICAL TRIAL: NCT00388869
Title: Calcifications of the Renal Arteries and Renal Artery Stenosis in Patients With and Without Hypertension?
Brief Title: Renal Artery Calcium and Hypertension
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: HILLER-HMO-CTIL
Record Dates: First submitted 2006-10-15; First posted 2006-10-17 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-10

CONDITIONS: Hypertension; Atherosclerosis
Keywords: renal artery; calcium; CT; hypertension
MeSH Terms: conditions — Hypertension; Atherosclerosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
CT of the abdomen is a very common examination performed for various indications.One of the common findings is vascular calcifications including calcifications of the renal arteries.Calcifications in the carotid arteries and coronary arteries are good predictor for obstructive atherosclerotic disease.Stenosis of the renal arteries can cause symptomatic or asymptomatic hypertension with subsequent clinical sequelae. Therefore early diagnosis of this condition is imperative.

The goal of our study is to investigate the correlation between incidental calcifications of the renal arteries in CT examinations and the presence of actual stenosis of these vessels in patients with and without hypertension.

DETAILED DESCRIPTION:
Every patient aged 30-100 referred for abdominal CT examination with IV contrast injection will be included in this study (total 300 patients.Prior to the examination relevant clinical data including history of hypertension and predisposing conditions for atherosclerotic disease, will be investigated. The patient will undergo conventional CT with no special procedures. The images will be review by the radiologist for the presence of renal arteries calcifications, renal arteries stenosis,plaque location, plaque burden and characterization and secondary renal pathology.

This study will not change the examination technique and is not associated with any inconvenience to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Every patient referred fo abdominal CT aged 30-100

Exclusion Criteria:

* Contraindication for IV contrast injection failure to demonstrate renal arteries with contrast refusal to sign an informed consent

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Nurith Hiller, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel